CLINICAL TRIAL: NCT04871711
Title: A Phase 3 Clinical Trial to Confirm Efficacy and Evaluate Safety of Twice-daily Delgocitinib Cream 20 mg/g Compared With Cream Vehicle for a 16-week Treatment Period in Adult Subjects With Moderate to Severe Chronic Hand Eczema (DELTA 1)
Brief Title: Efficacy and Safety of Delgocitinib Cream in Adults With Moderate to Severe Chronic Hand Eczema
Acronym: DELTA 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0133-1401; 2020-002960-30 (EudraCT Number); U1111-1284-2099 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-05

CONDITIONS: Chronic Hand Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delgocitinib cream 20 mg/g (Experimental): Twice-daily topical application for 16 weeks
  Interventions: Drug: Delgocitinib cream
- Cream vehicle (Placebo Comparator): Twice-daily topical application for 16 weeks
  Interventions: Drug: Cream vehicle

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application
  Other Names: LEO 124249 cream
  Arms: Delgocitinib cream 20 mg/g
Drug: Cream vehicle — The cream vehicle is similar to the delgocitinib cream> except that it does not contain any active ingredient.
  Arms: Cream vehicle

SUMMARY:
This was a 16-week study in adult participants with chronic hand eczema (CHE). > The participants visited the clinic regularly to have the study doctor assess their CHE and to answer questions about itch, pain, CHE symptoms, and quality of life.

> The purpose was to assess how delgocitinib cream works to treat CHE when compared to a placebo cream with no active substance.

ELIGIBILITY:
Main inclusion criteria:

* Diagnosis of CHE, defined as hand eczema that has persisted for more than 3 months or returned twice or more within the last 12 months.
* Disease severity graded as moderate to severe at screening and baseline according to Investigator's Global Assessment for chronic hand eczema (IGA-CHE) (i.e. an IGA-CHE score of 3 or 4).
* Hand Eczema Symptom Diary (HESD) itch score (weekly average) of ≥4 points at baseline.
* Participants who have a documented recent history of inadequate response to treatment with topical corticosteroids (TCS) or for whom TCS are documented to be otherwise medically inadvisable (e.g. due to important side effects or safety risks).
* Participants adherent to standard non-medicated skin care including avoidance of known and relevant irritants and allergens.

Main exclusion criteria:

* Concurrent skin diseases on the hands, e.g. tinea manuum.
* Active atopic dermatitis requiring medical treatment in regions other than the hands and feet.
* Active psoriasis on any part of the body.
* Hyperkeratotic hand eczema in combination with a history of psoriasis on any part of the body.
* Clinically significant infection on the hands.
* Systemic treatment with immunosuppressive drugs, immunomodulating drugs, retinoids, or corticosteroids within 28 days prior to baseline.
* Use of tanning beds, phototherapy, or bleach baths on the hands within 28 days prior to baseline.
* Previous or current treatment with Janus kinase (JAK) inhibitors (including delgocitinib/LEO 124249), systemic or topical.
* Cutaneously applied treatment with immunomodulators or TCS on the hands within 14 days prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 14 days prior to baseline.
* Other transdermal or cutaneously applied therapy on the hands (except for the use of subject's own emollients) within 7 days prior to baseline.
* Cutaneously applied treatments in regions other than the hands, which could interfere with clinical trial evaluations or pose a safety concern within 7 days prior to baseline.
* Treatment with any marketed biological therapy or investigational biologic agents:

  * Any cell-depleting agents: within 6 months prior to baseline, or until lymphocyte count returns to normal, whichever is longer.
  * Other biologics: within 3 months or 5 half-lives, whichever is longer, prior to baseline.
* Clinically significant infection within 28 days prior to baseline which, in the opinion of the investigator, may compromise the safety of the participant in the trial, interfere with evaluation of the IMP, or reduce the participant's ability to participate in the trial.
* History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the participant taking antiretroviral medications as determined by medical history and/or participant's verbal report.
* Any disorder which is not stable and could:

  * Affect the safety of the participant throughout the trial.
  * Impede the participant's ability to complete the trial.
* Positive hepatitis B surface antigen or hepatitis C virus antibody serology at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (50):
- Canada (8):
  - LEO Investigational Site, Calgary, Alberta
  - LEO Investigational Site, Edmonton, Alberta
  - LEO Investigational Site, Red Deer, Alberta
  - LEO Investigational Site, Kingston, Ontario
  - LEO Investigational Site, London, Ontario
  - LEO Investigational Site, Markham, Ontario
  - LEO Investigational Site, Toronto, Ontario
  - LEO Investigational Site, Montreal, Quebec
- France (13):
  - LEO Investigational Site, Nice, Alpes-Maritimes
  - LEO Investigational Site, Reims, Ardennes
  - LEO Investigational Site, Nantes, Loire-Atlantique 6
  - LEO Investigational Site, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - LEO Investigational Site, Lille, Nord
  - LEO Investigational Site, Le Mans, Sarthe
  - LEO Investigational Site, Bordeaux
  - LEO Investigational Site, Dijon
  - LEO Investigational Site, Lorient
  - LEO Investigational Site, Martigues
  - LEO Investigational Site, Nice
  - LEO Investigational Site, Paris
  - LEO Investigational Site, Toulouse
- Germany (10):
  - LEO Investigational Site, Berlin
  - LEO Investigational Site, Dresden
  - LEO Investigational Site, Gera
  - LEO Investigational Site, Göttingen
  - LEO Investigational Site, Hamburg
  - LEO Investigational Site, Haßfurt
  - LEO Investigational Site, Mainz
  - LEO Investigational Site, Memmingen
  - LEO Investigational Site, München
  - LEO Investigational Site, Osnabrück
- Italy (6):
  - LEO Investigational Site, Brescia
  - LEO Investigational Site, L’Aquila
  - LEO Investigational Site, Milan
  - LEO Investigational Site, Perugia
  - LEO Investigational Site, Roma
  - LEO Investigational Site, Vicenza
- Poland (7):
  - LEO Investigational Site, Bialystok
  - LEO Investigational Site, Gdansk
  - LEO Investigational Site, Krakow
  - LEO Investigational Site, Lodz
  - LEO Investigational Site, Lublin
  - LEO Investigational Site, Osielsko
  - LEO Investigational Site, Warsaw
- United Kingdom (6):
  - LEO Investigational Site, Salford, Greater Manchester
  - LEO Investigational Site, Leicester, Leicestershire
  - LEO Investigational Site, London, Leytonstone
  - LEO Investigational Site, Middlesbrough, North Yorkshire
  - LEO Investigational Site, Redhill, Surrey
  - LEO Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bissonnette R, Warren RB, Pinter A, Agner T, Gooderham M, Schuttelaar MLA, Crepy MN, Stingeni L, Serra-Baldrich E, Baranowski K, Korn S, Kurvits M, Plohberger U, Strange Vest N, Schliemann S; trial investigators. Efficacy and safety of delgocitinib cream in adults with moderate to severe chronic hand eczema (DELTA 1 and DELTA 2): results from multicentre, randomised, controlled, double-blind, phase 3 trials. Lancet. 2024 Aug 3;404(10451):461-473. doi: 10.1016/S0140-6736(24)01027-4. Epub 2024 Jul 18. PMID 39033766
- [Derived] Cohen D, Bewley A, Wollenberg A, Hong HC, Armstrong A, Jonsen E, Maslin D, Thoning H, von Eyben R, Chovatiya R. Matching-Adjusted Indirect Comparison of the Efficacy of Delgocitinib Cream and Dupilumab in the Treatment of Moderate to Severe Atopic Hand Eczema. Dermatol Ther (Heidelb). 2025 Nov 15. doi: 10.1007/s13555-025-01592-y. Online ahead of print. PMID 41240207
- [Derived] Silverberg JI, Agner T, Baranowski K, Plohberger U, Thoning H, Arbuckle R, Grant L, Skingley G, Bissonnette R. Validation of the Investigator Global Assessment of Chronic Hand Eczema (IGA-CHE): a new clinician reported outcome measure of CHE severity. Arch Dermatol Res. 2024 Mar 20;316(4):110. doi: 10.1007/s00403-024-02818-3. PMID 38507100
- [Derived] Molin S, Larsen LS, Joensson P, Oesterdal ML, Arbuckle R, Grant L, Skingley G, Schuttelaar MLA. Development and Psychometric Validation of a Patient-Reported Outcome Measure to Assess the Signs and Symptoms of Chronic Hand Eczema: The Hand Eczema Symptom Diary (HESD). Dermatol Ther (Heidelb). 2024 Mar;14(3):643-669. doi: 10.1007/s13555-024-01114-2. Epub 2024 Mar 15. PMID 38485862

RESULTS

PARTICIPANT FLOW:
Groups:
- Delgocitinib Cream 20 mg/g: Twice-daily topical application for 16 weeks >
  > Delgocitinib cream: Cream for topical application
- Cream Vehicle: Twice-daily topical application for 16 weeks >
  > Cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
Period: Overall Study
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Started | 325 | 162
Completed | 305 | 141
Not Completed | 20 | 21
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Lack of Efficacy | 5 | 7
Not completed — Adverse Event | 2 | 6
Not completed — Various reasons | 2 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Delgocitinib Cream 20 mg/g: Twice-daily topical application for 16 weeks>
  > Delgocitinib cream: Cream for topical application
- Cream Vehicle: Twice-daily topical application for 16 weeks>
  > Cream vehicle: The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
- Total: Total of all reporting groups
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle | Total
Number analyzed (Participants) | 325 | 162 | 487
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 297 | 154 | 451
  >=65 years | 28 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (14.3) | 42.9 (14.1) | 43.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 104 | 306
  Male | 123 | 58 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 4 | 18
  Not Hispanic or Latino | 292 | 147 | 439
  Unknown or Not Reported | 19 | 11 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 14 | 5 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 283 | 144 | 427
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 22 | 11 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 65 | 32 | 97
  Poland | 70 | 35 | 105
  United Kingdom | 20 | 4 | 24
  Italy | 31 | 14 | 45
  France | 49 | 32 | 81
  Germany | 90 | 45 | 135
Baseline IGA-CHE score [Count of Participants; unit: Participants] — The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 218 | 109 | 327
    4 - Severe | 107 | 53 | 160
Baseline HECSI score [Mean (Standard Deviation); unit: units on a scale] — The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity.
  units on a scale | 77.6 (46.4) | 77.3 (53.6) | 77.5 (48.9)
Baseline HESD itch score (weekly average) [Mean (Standard Deviation); unit: units on a scale] — The Hand Eczema Symptom Diary (HESD) itch score is one component of the HESD eDiary. In the HESD eDiary, participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. Population: Data not available for 1 participant in the delgocitinib cream 20 mg/g group.
  units on a scale
    number analyzed (Participants) | 324 | 162 | 486
    (all) | 7.13 (1.64) | 7.23 (1.69) | 7.16 (1.66)
Baseline HESD pain score (weekly average) [Mean (Standard Deviation); unit: units on a scale] — The Hand Eczema Symptom Diary (HESD) pain score is one component of the HESD eDiary. In the HESD eDiary, participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. Population: Data not available for 1 participant in the delgocitinib cream 20 mg/g group.
  units on a scale
    number analyzed (Participants) | 324 | 162 | 486
    (all) | 6.83 (2.00) | 6.84 (2.03) | 6.83 (2.01)
Baseline HESD score (weekly average) [Mean (Standard Deviation); unit: units on a scale] — The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. The HESD score is derived as the average of the 6 signs and symptoms. Population: Data not available for 1 participant in the delgocitinib cream 20 mg/g group.
  units on a scale
    number analyzed (Participants) | 324 | 162 | 486
    (all) | 7.15 (1.66) | 7.16 (1.68) | 7.16 (1.67)
Baseline DLQI score [Mean (Standard Deviation); unit: units on a scale] — The Dermatology Life Quality Index (DLQI) is a validated questionnaire consisting of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week. The DLQI score is the sum of the 10 items (score ranging from 0 to 30); a high score is indicative of a poor quality of life. Population: Data not available for 4 participants each in the delgocitinib cream 20 mg/g group and in the cream vehicle group.
  units on a scale
    number analyzed (Participants) | 321 | 158 | 479
    (all) | 12.8 (6.0) | 12.9 (6.8) | 12.8 (6.3)
Baseline HEIS score [Mean (Standard Deviation); unit: units on a scale] — The Hand Eczema Impact Scale (HEIS) addresses 9 items within the following domains: Proximal Daily Activity Limitations (PDAL), embarrassment with the appearance of the hands, frustration with CHE, sleep, work, and physical functioning. Each item is scored on a 5-point scale ranging from 0 (not at all) to 4 (extremely). The HEIS score is the average of the 9 items. Population: Data not available for 4 participants each in the delgocitinib cream 20 mg/g group and in the cream vehicle group.
  units on a scale
    number analyzed (Participants) | 321 | 158 | 479
    (all) | 2.50 (0.77) | 2.49 (0.89) | 2.49 (0.81)
Baseline HEIS PDAL score [Mean (Standard Deviation); unit: units on a scale] — Proximal Daily Activity Limitations (PDAL) is one of the domain scores in Hand Eczema Impact Scale (HEIS) assessing the participant's perceived impact on their daily activities. Each item is scored on a 5-point scale ranging from 0 (not at all) to 4 (extremely). HEIS PDAL score is the average of the 3 items. Population: Data not available for 4 participants each in the delgocitinib cream 20 mg/g group and in the cream vehicle group.
  units on a scale
    number analyzed (Participants) | 321 | 158 | 479
    (all) | 2.57 (0.89) | 2.57 (0.94) | 2.57 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With IGA-CHE TS at Week 16
Description: The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Participants | 64 | 16
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; Based on the primary analysis of the primary estimand 'composite'. Subjects with missing data, subjects who received rescue treatment, or subjects who permanently discontinued IMP were considered non-responders; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — 5% significance level (two-sided); Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 9.8, 95% CI 2-sided [3.6 to 16.1] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

2. Secondary Outcome: Number of Participants With Reduction of HESD Itch Score (Weekly Average) of ≥4 Points From Baseline at Week 16
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. This endpoint will only assess the 'itch' component and will be evaluated among participants with a baseline HESD itch score (weekly average) ≥4 points.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 323 | 161
Participants | 152 | 37
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Evaluated at 5% significance level (two-sided) using hierarchical tests, alpha splitting and alpha recycling controlling overall type 1 error at 5% (two-sided); Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 24.1, 95% CI 2-sided [15.5 to 32.6] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

3. Secondary Outcome: Number of Participants With Reduction of HESD Score (Weekly Average) of ≥4 Points From Baseline at Week 16
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. The HESD score is derived as the average of the 6 signs and symptoms. This endpoint will be evaluated among participants with a baseline HESD score (weekly average) ≥4 points.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 309 | 156
Participants | 146 | 38
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 22.8, 95% CI 2-sided [14.0 to 31.7] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

4. Secondary Outcome: Number of Participants With IGA-CHE TS at Week 8
Description: The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global CHE and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Participants | 74 | 17
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Evaluated at 4% significance level (two-sided) using hierarchical tests, alpha splitting and alpha recycling controlling overall type 1 error at 5% (two-sided); Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 12.3, 95% CI 2-sided [5.7 to 18.9] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

5. Secondary Outcome: Number of Participants With IGA-CHE TS at Week 4
Description: as for outcome 4
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Participants | 50 | 8
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 10.4, 95% CI 2-sided [5.3 to 15.6] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

6. Secondary Outcome: Number of Participants With Reduction of HESD Itch Score (Weekly Average) of ≥4 Points From Baseline at Week 8
Description: as for outcome 2
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 323 | 161
Participants | 138 | 35
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 21.0, 95% CI 2-sided [12.6 to 29.4] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

7. Secondary Outcome: Number of Participants With Reduction of HESD Itch Score (Weekly Average) of ≥4 Points From Baseline at Week 4
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 323 | 161
Participants | 99 | 18
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 19.5, 95% CI 2-sided [12.5 to 26.5] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

8. Secondary Outcome: Number of Participants With Reduction of HESD Itch Score (Weekly Average) of ≥4 Points From Baseline at Week 2
Description: as for outcome 2
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 323 | 161
Participants | 50 | 10
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 9.3, 95% CI 2-sided [3.8 to 14.7] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

9. Secondary Outcome: Number of Participants With Reduction of HESD Score (Weekly Average) of ≥4 Points From Baseline at Week 8
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 309 | 156
Participants | 123 | 27
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 22.5, 95% CI 2-sided [14.4 to 30.6] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

10. Secondary Outcome: Number of Participants With Reduction of HESD Score (Weekly Average) of ≥4 Points From Baseline at Week 4
Description: as for outcome 3
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 309 | 156
Participants | 92 | 16
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 19.5, 95% CI 2-sided [12.5 to 26.5] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

11. Secondary Outcome: Number of Participants With Reduction of HESD Pain Score (Weekly Average) of ≥4 Points From Baseline at Week 16
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. This endpoint will only assess the 'pain' component and will be evaluated among participants with a baseline HESD pain score (weekly average) ≥4 points.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 291 | 149
Participants | 143 | 41
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 21.7, 95% CI 2-sided [12.4 to 30.9] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

12. Secondary Outcome: Number of Participants With Reduction of HESD Pain Score (Weekly Average) of ≥4 Points From Baseline at Week 8
Description: as for outcome 11
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 291 | 149
Participants | 134 | 33
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 23.9, 95% CI 2-sided [15.2 to 32.7] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

13. Secondary Outcome: Number of Participants With Reduction of HESD Pain Score (Weekly Average) of ≥4 Points From Baseline at Week 4
Description: as for outcome 11
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 291 | 149
Participants | 100 | 22
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 19.6, 95% CI 2-sided [11.8 to 27.5] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

14. Secondary Outcome: Number of Participants With HECSI-90 at Week 16
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity. HECSI-90 is defined as at least 90% improvement in HECSI score from baseline.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Participants | 96 | 20
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Evaluated at 1% significance level (two-sided) using hierarchical tests, alpha splitting and alpha recycling controlling overall type 1 error at 5% (two-sided); Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 17.2, 95% CI 2-sided [10.1 to 24.3] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

15. Secondary Outcome: Number of Participants With HECSI-75 at Week 16
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity. HECSI-75 is defined as at least 75% improvement in HECSI score from baseline.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Participants | 160 | 38
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 14, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 25.7, 95% CI 2-sided [17.2 to 34.3] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

16. Secondary Outcome: Number of Participants With HECSI-75 at Week 8
Description: as for outcome 15
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Participants | 163 | 42
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 14, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 24.2, 95% CI 2-sided [15.5 to 33.0] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

17. Secondary Outcome: Percentage Change in HECSI Score From Baseline to Week 16
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
percentage change | -56.5 (3.4) | -21.2 (4.8)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; Primary analysis of primary estimand 'composite'. Missing data for subjects who did not attend the visit was imputed as WOCF (including baseline value). For subjects who received rescue treatment or subjects who have permanently discontinued the IMP, observed data was considered non-response by using WOCF (including baseline value); Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline HECSI score; Mean Difference (Net) = -35.2, 95% CI 2-sided [-46.7 to -23.8]

18. Secondary Outcome: Change in DLQI Score From Baseline to Week 16
Description: The Dermatology Life Quality Index (DLQI) is a validated questionnaire consisting of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week. The DLQI score is the sum of the 10 items (score ranging from 0 to 30); a high score is indicative of a poor quality of life.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 321 | 158
score on a scale | -7.6 (0.3) | -3.9 (0.4)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline DLQI score; Mean Difference (Net) = -3.6, 95% CI 2-sided [-4.7 to -2.6]

19. Secondary Outcome: Change in HESD Score (Weekly Average) From Baseline to Week 16
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. The HESD score is derived as the average of the 6 signs and symptoms.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 324 | 162
score on a scale | -3.4 (0.1) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline HESD score; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.2 to -1.2]

20. Secondary Outcome: Change in HESD Itch Score (Weekly Average) From Baseline to Week 16
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. This endpoint will only assess the 'itch' component.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 324 | 162
score on a scale | -3.6 (0.2) | -1.9 (0.2)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline HESD itch score; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.3 to -1.2]

21. Secondary Outcome: Change in HESD Pain Score (Weekly Average) From Baseline to Week 16
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. This endpoint will only assess the 'pain' component.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 324 | 162
score on a scale | -3.4 (0.2) | -1.8 (0.2)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline HESD pain score; Mean Difference (Net) = -1.6, 95% CI 2-sided [-2.1 to -1.0]

22. Secondary Outcome: Change in HEIS Score From Baseline to Week 16
Description: The Hand Eczema Impact Scale (HEIS) addresses 9 items within the following domains: Proximal Daily Activity Limitations (PDAL), embarrassment with the appearance of the hands, frustration with CHE, sleep, work, and physical functioning. Each item is scored on a 5-point scale ranging from 0 (not at all) to 4 (extremely). The HEIS score is the average of the 9 items.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 321 | 158
score on a scale | -1.46 (0.05) | -0.82 (0.08)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline HEIS score; Mean Difference (Net) = -0.64, 95% CI 2-sided [-0.83 to -0.45]

23. Secondary Outcome: Change in HEIS PDAL Score From Baseline to Week 16
Description: Proximal Daily Activity Limitations (PDAL) is one of the domain scores in Hand Eczema Impact Scale (HEIS) assessing the participant's perceived impact on their daily activities. Each item is scored on a 5-point scale ranging from 0 (not at all) to 4 (extremely). HEIS PDAL score is the average of the 3 items.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 321 | 158
score on a scale | -1.46 (0.06) | -0.86 (0.08)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; Adjusted for treatment, region, baseline IGA-CHE score, and baseline HEIS PDAL score; Mean Difference (Net) = -0.6, 95% CI 2-sided [-0.79 to -0.40]

24. Secondary Outcome: Reduction of DLQI Score of ≥4 Points From Baseline at Week 16
Description: The Dermatology Life Quality Index (DLQI) is a validated questionnaire consisting of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week. The DLQI score is the sum of the 10 items (score ranging from 0 to 30); a high score is indicative of a poor quality of life. This endpoint will be evaluated among participants with a baseline DLQI score ≥4 points.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 305 | 148
Participants | 227 | 74
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Cream Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 14, analysis 1]; Stratified by region and baseline IGA-CHE score; Risk Difference (RD) = 24.5, 95% CI 2-sided [15.0 to 33.9] — Mantel-Haenszel risk difference, stratified by region and baseline IGA-CHE score

25. Secondary Outcome: Number of Treatment-emergent AEs From Baseline up to End of Trial
Description: An adverse event (AE) were considered treatment emergent if started after the first application of investigational medicinal product (IMP), or if started before the first application of IMP and worsened in severity after first dose of IMP. End of trial was defined as Week 16 for participants who rolled over to the long-term extension trial and as Week 18 for participants who did not roll over.
Time Frame: 16 weeks (18 weeks for participants not participating in the long-term extension trial [LP0133-1403])
Measure: Number; unit: Adverse events
Arm/Group | Delgocitinib Cream 20 mg/g | Cream Vehicle
Number analyzed (Participants) | 325 | 162
Adverse events | 308 | 161

ADVERSE EVENTS:
Time Frame: 16 weeks (18 weeks for participants not participating in the long-term extension trial [LP0133-1403])
Groups:
- Delgocitinib |20 mg/g; Vehicle|: Twice-daily topical application for 16 weeks
Arm/Group | Delgocitinib |20 mg/g | Vehicle|
All-Cause Mortality (participants affected / at risk) | 0/325 | 0/162
Serious Adverse Events (participants affected / at risk) | 6/325 | 3/162
Other Adverse Events (participants affected / at risk) | 69/325 | 42/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib |20 mg/g (N=325) | Vehicle| (N=162)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Keratitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib |20 mg/g (N=325) | Vehicle| (N=162)
Allergy to metals (Immune system disorders) | 7 (7) | 3 (3)
COVID-19 (Infections and infestations) | 35 (35) | 14 (14)
Nasopharyngitis (Infections and infestations) | 23 (25) | 14 (16)
Headache (Nervous system disorders) | 9 (13) | 4 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma seeks publication of all Phase 3 clinical trials in peer-reviewed journals within 18 months of trial completion, regardless of whether the findings are positive or negative. If there is no multi-center publication within 18 months after the clinical trial has been completed or terminated at all trial sites, the investigator has the right to publish the results from the clinical trial generated by the investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04871711/Prot_SAP_000.pdf